CLINICAL TRIAL: NCT04805229
Title: Using Difference-in-Differences to Evaluate the Effect of a Statewide Quality Improvement Program on New Persistent Opioid Use After Surgery
Brief Title: A Difference-In-Differences Analysis of New Persistent Opioid Use After Surgery
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Chad Brummett, Professor of Anesthesiology, University of Michigan
Other Study IDs: HUM00119139
Record Dates: First submitted 2021-03-15; First posted 2021-03-18 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2020-10

CONDITIONS: Opioid Use

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing surgery: Retrospective cohort of patients who underwent surgery between 1/1/13 to 12/31/19 and were sampled from the Truven Health MarketScan Database.
  Interventions: Other: Retrospective analysis of opioid use after surgery

INTERVENTIONS:
Other: Retrospective analysis of opioid use after surgery — Retrospective analysis of opioid use after one of the following surgical procedure categories: laparoscopic cholecystectomy, laparoscopic appendectomy, minor hernia repair (including laparoscopic or open inguinal, femoral, umbilical, and epigastric hernia repair), open and laparoscopic ventral/incisional hernia repair, laparoscopic colectomy, open colectomy, vaginal hysterectomy, laparoscopic hysterectomy, and open abdominal hysterectomy.

SUMMARY:
The Michigan Opioid Prescribing and Engagement Network (M-OPEN) was established in 2016 with the goal of reducing excessive opioid prescribing after surgery using evidence-based prescribing guidelines. Beginning in July 2016, M-OPEN began a statewide quality improvement campaign to educate providers and share prescribing best practices. This retrospective study examines the effect of these efforts on new persistent opioid use after surgery compared to other states where no such program existed using a difference-in-differences approach.

DETAILED DESCRIPTION:
In the United States, surgical care has become a gateway for chronic opioid dependence and its associated morbidity. Between 5-10% of patients who receive opioids for postoperative pain control go on to develop long-term opioid use. This translates to more than 2 million previously opioid-naïve individuals developing chronic opioid use after surgery each year. Persistent opioid use after surgery is associated with increased readmissions, healthcare utilization, and healthcare expenditures. Critically, long-term opioid use increases the risk of overdose and death in patients who, prior to their surgery, had no exposure to opioids.

Growing recognition of this problem has led to numerous efforts aimed at reducing opioid-associated morbidity after surgery. These include legislative limits on opioid prescribing for acute pain, procedure-specific prescribing guidelines based on patient-reported opioid use, and opioid-sparing pain management pathways. In Michigan specifically, the Michigan Opioid Prescribing and Engagement Network (M-OPEN) led a statewide quality improvement effort beginning in 2016 that focused on provider education using evidence-based opioid prescribing guidelines. Previously, these guidelines have been shown to significantly reduce excessive postoperative opioid prescribing across the state, however it is currently unknown whether these efforts have had any effect on the actual incidence of persistent opioid use after surgery.

Therefore, the current study will evaluate the incidence of new persistent opioid use before and after the establishment of M-OPEN in Michigan. Beginning in 2016, a statewide quality improvement initiative was undertaken in Michigan to improve postoperative opioid prescribing. In order to accomplish this goal, this study will use a difference-in-differences approach to compare new persistent opioid use in Michigan before and after 2016 to other states where no such quality improvement effort existed.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 years and older)
* Patients undergoing one of the following procedures: laparoscopic cholecystectomy, laparoscopic appendectomy, minor hernia repair (including laparoscopic or open inguinal, femoral, umbilical, and epigastric hernia repair), open and laparoscopic ventral/incisional hernia repair, laparoscopic colectomy, open colectomy, vaginal hysterectomy, laparoscopic hysterectomy, and open abdominal hysterectomy
* Patients who underwent surgery between January 1, 2013 and December 31, 2019

Exclusion Criteria:

* Patients who are not opioid-naive at the time of surgery, defined as filling 1 or more opioid prescriptions between the 12 months to 31 days prior to surgery
* Patients without continuous insurance enrollment for at least 12 months before and at least 6 months after the date of surgery
* Patients still in the hospital on postoperative day 30
* Patients not discharged home after surgery
* Patients who underwent another surgery within 6 months of their index operation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Data for this study will be obtained from the Truven Health MarketScan database, which is a national data set of employer-based insurance claims. Patients in the database who underwent one of the eligible procedures will be identified using Current Procedural Terminology codes that correspond to the specific operations under analysis.
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
The change in the incidence of new persistent opioid use before and after July 2016 in Michigan compared to all other states. | Postoperative days 4 to 180
  Among patients who undergo surgery, new persistent opioid use is defined as filling an opioid prescription in post-discharge days 4-90 and filling another opioid prescription in post-discharge days 91-180. This incidence will be measured from 1/1/13-6/30/16 (before M-OPEN established) and from 7/1/16-12/31/19 (after M-OPEN established) and the change before and after this date will be compared between Michigan and all other states (the difference-in-differences). Outcomes will be measured at 1 year, 2 years, and 3 years post-intervention.

SECONDARY OUTCOMES:
The change in the incidence of new persistent opioid use before and after July 2016 in Michigan compared to Indiana and Wisconsin | Postoperative days 4 to 180
  Among patients who undergo surgery, new persistent opioid use is defined as filling an opioid prescription in post-discharge days 4-90 and filling another opioid prescription in post-discharge days 91-180. This incidence will be measured from 1/1/13-6/30/16 (before M-OPEN established) and from 7/1/16-12/31/19 (after M-OPEN established) and the change before and after this date will be compared between Michigan and Indiana/Wisconsin (the difference-in-differences). Outcomes will be measured at 1 year, 2 years, and 3 years post-intervention.
The change in the incidence of new persistent opioid use before and after July 2016 in Michigan compared to 11 other Midwest states (Illinois, Indiana, Iowa, Kansas, Minnesota, Missouri, Nebraska, North Dakota, Ohio, South Dakota, and Wisconsin). | Postoperative days 4 to 180
  Among patients who undergo surgery, new persistent opioid use is defined as filling an opioid prescription in post-discharge days 4-90 and filling another opioid prescription in post-discharge days 91-180. This incidence will be measured from 1/1/13-6/30/16 (before M-OPEN established) and from 7/1/16-12/31/19 (after M-OPEN established) and the change before and after this date will be compared between Michigan and 11 other Midwest states. Outcomes will be measured at 1 year, 2 years, and 3 years post-intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Chad Brummett, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Waljee JF, Li L, Brummett CM, Englesbe MJ. Iatrogenic Opioid Dependence in the United States: Are Surgeons the Gatekeepers? Ann Surg. 2017 Apr;265(4):728-730. doi: 10.1097/SLA.0000000000001904. No abstract available. PMID 27429023
- [Background] Hah JM, Bateman BT, Ratliff J, Curtin C, Sun E. Chronic Opioid Use After Surgery: Implications for Perioperative Management in the Face of the Opioid Epidemic. Anesth Analg. 2017 Nov;125(5):1733-1740. doi: 10.1213/ANE.0000000000002458. PMID 29049117
- [Background] Brummett CM, Waljee JF, Goesling J, Moser S, Lin P, Englesbe MJ, Bohnert ASB, Kheterpal S, Nallamothu BK. New Persistent Opioid Use After Minor and Major Surgical Procedures in US Adults. JAMA Surg. 2017 Jun 21;152(6):e170504. doi: 10.1001/jamasurg.2017.0504. Epub 2017 Jun 21. PMID 28403427
- [Background] Lee JS, Hu HM, Edelman AL, Brummett CM, Englesbe MJ, Waljee JF, Smerage JB, Griggs JJ, Nathan H, Jeruss JS, Dossett LA. New Persistent Opioid Use Among Patients With Cancer After Curative-Intent Surgery. J Clin Oncol. 2017 Dec 20;35(36):4042-4049. doi: 10.1200/JCO.2017.74.1363. Epub 2017 Oct 19. PMID 29048972
- [Background] Harbaugh CM, Lee JS, Hu HM, McCabe SE, Voepel-Lewis T, Englesbe MJ, Brummett CM, Waljee JF. Persistent Opioid Use Among Pediatric Patients After Surgery. Pediatrics. 2018 Jan;141(1):e20172439. doi: 10.1542/peds.2017-2439. Epub 2017 Dec 4. PMID 29203521
- [Background] Brescia AA, Waljee JF, Hu HM, Englesbe MJ, Brummett CM, Lagisetty PA, Lagisetty KH. Impact of Prescribing on New Persistent Opioid Use After Cardiothoracic Surgery. Ann Thorac Surg. 2019 Oct;108(4):1107-1113. doi: 10.1016/j.athoracsur.2019.06.019. Epub 2019 Aug 22. PMID 31447051
- [Background] Lee JS, Vu JV, Edelman AL, Gunaseelan V, Brummett CM, Englesbe MJ, Waljee JF. Health Care Spending and New Persistent Opioid Use After Surgery. Ann Surg. 2020 Jul;272(1):99-104. doi: 10.1097/SLA.0000000000003399. PMID 31851641
- [Background] Babu KM, Brent J, Juurlink DN. Prevention of Opioid Overdose. N Engl J Med. 2019 Jun 6;380(23):2246-2255. doi: 10.1056/NEJMra1807054. No abstract available. PMID 31167053
- [Background] Howard R, Waljee J, Brummett C, Englesbe M, Lee J. Reduction in Opioid Prescribing Through Evidence-Based Prescribing Guidelines. JAMA Surg. 2018 Mar 1;153(3):285-287. doi: 10.1001/jamasurg.2017.4436. PMID 29214318
- [Background] Overton HN, Hanna MN, Bruhn WE, Hutfless S, Bicket MC, Makary MA; Opioids After Surgery Workgroup. Opioid-Prescribing Guidelines for Common Surgical Procedures: An Expert Panel Consensus. J Am Coll Surg. 2018 Oct;227(4):411-418. doi: 10.1016/j.jamcollsurg.2018.07.659. Epub 2018 Aug 14. PMID 30118896
- [Background] Hallway A, Vu J, Lee J, Palazzolo W, Waljee J, Brummett C, Englesbe M, Howard R. Patient Satisfaction and Pain Control Using an Opioid-Sparing Postoperative Pathway. J Am Coll Surg. 2019 Sep;229(3):316-322. doi: 10.1016/j.jamcollsurg.2019.04.020. Epub 2019 May 30. PMID 31154092
- [Background] Vu JV, Howard RA, Gunaseelan V, Brummett CM, Waljee JF, Englesbe MJ. Statewide Implementation of Postoperative Opioid Prescribing Guidelines. N Engl J Med. 2019 Aug 15;381(7):680-682. doi: 10.1056/NEJMc1905045. No abstract available. PMID 31412184
- [Background] Brown CS, Vu JV, Howard RA, Gunaseelan V, Brummett CM, Waljee J, Englesbe M. Assessment of a quality improvement intervention to decrease opioid prescribing in a regional health system. BMJ Qual Saf. 2021 Mar;30(3):251-259. doi: 10.1136/bmjqs-2020-011295. Epub 2020 Sep 16. PMID 32938775
- [Background] Hill MV, Stucke RS, Billmeier SE, Kelly JL, Barth RJ Jr. Guideline for Discharge Opioid Prescriptions after Inpatient General Surgical Procedures. J Am Coll Surg. 2018 Jun;226(6):996-1003. doi: 10.1016/j.jamcollsurg.2017.10.012. Epub 2017 Nov 30. PMID 29198638